CLINICAL TRIAL: NCT07277296
Title: A Multicenter, Single-arm, Pivotal Study to Evaluate the Safety and Efficacy of the SwitchGuard™ Neuroprotection System (NPS) for Providing Cerebral Embolic Protection During Carotid Artery Stenting Via the Transcarotid Artery Revascularization (TCAR) Approach When Used in Conjunction With the CGuard™ Prime 80 Carotid Stent System
Brief Title: CGUARDIANS III IDE Pivotal Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InspireMD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGUARDIANS III
Record Dates: First submitted 2025-12-02; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Carotid Artery Stenosis
Keywords: Transcarotid Artery Revascularization; Carotid Endarterectomy
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Experimental): SwitchGuardTM NPS
  Interventions: Device: SwitchGuardTM NPS

INTERVENTIONS:
Device: SwitchGuardTM NPS — The CGuard Prime™ 80 will be used in conjunction with the SwitchGuard™ NPS for the carotid artery stenting implantation procedure that will be performed by physician investigators experienced with transcarotid artery revascularization.

SUMMARY:
This is a prospective, multi-center, single-arm, pivotal study. The objective of this study is to evaluate the safety and efficacy of the SwitchGuard NPS in providing cerebral embolic protection during Transcarotid Artery Revascularization procedures using the CGuard Prime Carotid Stent System 80 in the treatment of carotid artery stenosis in patients at high risk for complications from CEA.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, single arm pivotal study. The study shall not be blinded prior to, during or following the procedure. Patients undergoing transcarotid artery revascularization will be screened against the study inclusion/exclusion criteria. If the patient meets study eligibility requirements, they shall be invited to participate, provided informed consent and shall subsequently be assigned a study ID number.

Enrollment will be 103 pivotal patients. A maximum of 20% of patients will be enrolled at any single site. The total enrollment accounts for an estimate that up to 2 patients will exit the study prior to the 30-day primary endpoint assessment.

An additional roll-in cohort of up to 2 patients per primary physician operator at each study site may also be accrued (maximum of 50 roll-in patients total, assuming one primary physician operator per site).

This study does not duplicate any current knowledge existing today on use of the SwitchGuard NPS when used in conjunction with the CGuard Prime™ 80cm in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing and able to provide appropriate study-specific informed consent, follow protocol procedures, and comply with follow-up visit requirements.
2. Patient is diagnosed with carotid artery disease treatable with a Carotid Artery Stent via a Transcarotid Artery Revascularization approach and is either symptomatic or asymptomatic, defined as:

   Symptomatic carotid stenosis ≥ 50%. Symptomatic is defined as amaurosis fugax, transient ischemia attack (TIA) or stroke within the last 6 months ipsilateral to the side of the stenosis OR asymptomatic carotid stenosis ≥ 80%
3. High Risk condition for CEA: at least one, as shown below:

Comorbid conditions:

Age ≥ 70 (maximum 82 years) CCS angina class 3-4 or unstable angina Congestive Heart Failure (CHF) NYHA class III-IV Left ventricular ejection fraction (LVEF) ≤ 35% MI ≥ 72 hours and < 6 weeks pre-procedure Multi-vessel CAD (≥ 2 vessels >70% stenosis) and history of angina Chronic Obstructive Pulmonary Disease (COPD) with FEV1<50 Permanent contralateral cranial nerve injury/paralysis Restenosis from previous carotid endarterectomy (CEA) Planned coronary artery bypass grafting (CABG) or valve replacement surgery between 31-60 days after CAS Abdominal aortic aneurysm surgical repair or Endovascular repair is planned between 31 to 60 days after CAS

Anatomic conditions:

Occlusion of the contralateral CCA or ICA Prior radiation treatment to the neck or a radical neck dissection Severe bilateral ICA stenosis requiring treatment Target lesion at or above the level of the jaw (C2) or below the clavicle Severe tandem lesions Inability to extend the neck due to cervical disorders Laryngeal palsy or laryngectomy Prior head and neck surgery in the region of the carotid artery Tracheostomy or tracheostoma Spinal immobility of the neck

Exclusion Criteria:

1. Patient had or will have an interventional procedure or surgery of the carotid, coronary or peripheral arteries within 30 days before or after the index carotid procedure
2. Patient had or will have open heart surgery or valvular intervention (percutaneous or surgical), or any major operation, within 30 days before or after the index carotid procedure
3. Vascular anatomy that would preclude safe sheath insertion or deliverability of stent
4. Previously placed stent in the ipsilateral ICA or CCA
5. Total occlusion or presence of a "string sign" of the ipsilateral ICA or CCA
6. Presence of a filling defect of the target lesion
7. Tandem lesions, which cannot be covered by a single CGuard Prime stent
8. Stenosis of the innominate artery or proximal CCA requiring revascularization
9. Open neck stoma
10. History of bleeding diatheses or coagulopathy
11. Hypercoagulable state
12. Alternative source of cerebral embolus, including but not limited to:

Chronic atrial fibrillation Episode(s) of paroxysmal atrial fibrillation within the past 6 months or history of paroxysmal atrial fibrillation requiring chronic anticoagulation Knowledge of cardiac sources of embolus (e.g. left ventricular aneurysm, intracardiac filling defect, cardiomyopathy, aortic or mitral prosthetic heart valve, calcific aortic stenosis, endocarditis, mitral stenosis, atrial septal defect, atrial septal aneurysm, or left atrial myxoma) Recently (<60 days) implanted heart valve (either surgically or endovascularly) as a known source of emboli as confirmed on echocardiogram, Abnormal angiographic findings: ipsilateral intracranial or extracranial arterial stenosis (as determined by angiography or CTA/MRA 6 months prior to index procedure) greater in severity than the lesion to be treated; cerebral aneurysm > 5mm; AVM (arteriovenous malformation) of the cerebral vasculature, or other abnormal angiographic findings Known sensitivity or allergy to nickel or titanium.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Composite primary endpoint | 30 days
  Incidence of the composite primary endpoint comprised of Death (all-cause mortality), all Stroke, or Myocardial Infarction (DSMI) through 30-days post-index procedure, based on Clinical Events Committee (CEC) adjudication.

SECONDARY OUTCOMES:
Rate of all death within 30 days of the procedure | 30 days
Rate of cardiac death within 30 days of the index procedure | 30 days
Rate of neurological death within 30 days of the index procedure | 30 days
Rate of all strokes within 30 days of the procedure | 30 days
Rate of major stroke within 30 days of the procedure | 30 days
Rate of minor stroke within 30 days of the procedure | 30 days
Rate of ipsilateral stroke within 30 days of the procedure | 30 days
Rate of MI within 30 days of the procedure | 30 days
Composite of death or stroke rate within 30 days of the procedure | 30 days
Rate of cranial nerve injury within 30 days of the procedure | 30 days
Access site complications (arterial/venous) | At procedure
All device-related serious adverse events within 30 days of the procedure | 30 days
Acute success for the SwitchGuard NPS | At procedure
  Successful insertion of the SwitchGuard NPS into the vasculature, followed by flow reversal, and the removal of the SwitchGuard NPS from the vasculature.
Acute success for CGuard Prime 80cm Delivery System and Stent | At procedure
  Successful insertion of the delivery system, successful deployment of the stent, and successful retraction of the delivery system when used in conjunction with the SwitchGuard NPS.
Technical Success for the CGuard Prime 80cm Delivery System and Stent | At procedure
  Technical Success Rate is defined as the number of patients with at least one CGuard Prime™ 80 device successfully delivered and deployed with final residual diameter stenosis < 30% following final post-balloon dilatation (if performed) divided by the total number of patients where CGuard Prime™ 80 device deployment was attempted when used in conjunction with the SwitchGuard NPS during a TCAR procedure.
Procedural success | 30 days
  Acute device success for CGuard Prime 80cm Delivery System and Stent, AND acute device success for SwitchGuard NPS, AND freedom from the composite of death, all stroke or MI at 30-day post-procedure.
Treatment Success for the CGuard Prime 80cm Delivery System and Stent | 30 days
  Treatment Success Rate is defined as the number of patients who meet CGuard Prime™ 80 Technical Success Rate without experiencing death, stroke or MI through 30-day post-procedure, divided by the total number of patients where CGuard Prime™ 80 device deployment was attempted when used in conjunction with the SwitchGuard NPS during a TCAR procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Geraghty, MD, Principal Investigator — Washington University School of Medicine; Patrick Edward Muck, MD, Principal Investigator — TriHealth Inc.